CLINICAL TRIAL: NCT04637698
Title: Phase Ib/II Study of OH2 Injection, an Oncolytic Type 2 Herpes Simplex Virus Expressing Granulocyte Macrophage Colony-Stimulating Factor, in Pancreatic Cancer
Brief Title: OH2 Oncolytic Viral Therapy in Pancreatic Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Strategy adjustment
Sponsor: Binhui Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BH-OH2-006
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Pancreatic Cancer
Keywords: Oncolytic Virus
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose expansion (Experimental): OH2 injection will be administered at 1E+07 CCID50/mL .
  Interventions: Biological: OH2 injection

INTERVENTIONS:
Biological: OH2 injection — Oncolytic Type 2 Herpes Simplex Virus

SUMMARY:
This phase Ib/II study evaluates the safety and efficacy of OH2 in patients with locally advanced/metastatic pancreatic cancer who have failed first-line standard treatment.

OH2 is an oncolytic virus developed upon genetic modifications of the herpes simplex virus type 2 strain HG52, allowing the virus to selectively replicate in tumors. Meanwhile, the delivery of the gene encoding human granulocyte macrophage colony-stimulating factor (GM-CSF) may induce a more potent antitumor immune response.

DETAILED DESCRIPTION:
OH2 injection ≤ 4 mL, administered by intratumoral injection of EUS-FNA, administered on the first day of the first cycle, every 3 weeks thereafter, administered on the 1st day of each cycle ± 3 days, continuous administration does not more than 6 treatment cycles.

ELIGIBILITY:
Inclusion Criteria:

1. The non-operative stage III or stage IV locally advanced or metastatic pancreatic cancer patients with clear diagnosis by pathology and/ or cytology.
2. Life expectancy >3 months.
3. Have received at least first-line or more systemic chemotherapy and failed. The definition of failure: Receiving first-line systemic chemotherapy means having used first-line chemotherapy such as gemcitabine, or tigeo capsule, or albumin paclitaxel, or liposomal irinotecan, or FOLFINOX.During or after treatment, the disease progression or toxic side effects are intolerable, and there must be imaging evidence or clinical evidence to prove the disease progression. For neoadjuvant/adjuvant therapy (chemotherapy or radiotherapy), if disease progression occurs during treatment or within 6 months after stopping treatment, it should be counted as a failure of first-line treatment;
4. Prior anti-tumor treatment including systemic, radical/extensive radiotherapy, targeted therapy, immunotherapy was over 28 days;
5. According to RECIST version 1.1, there is at least one measurable lesion that is suitable for intratumoral injection. The measured non-nodular lesions is defined as the longest diameter ≥ 10 mm . For lymph node lesions, the short diameter is ≥ 15 mm.If the measurable lesions located in the radiation field of previous radiotherapy or after local treatment are confirmed to have progressed, they can also be selected as target lesions.
6. General physical condition score ECOG 0 ≤ 2 (including boundary value);
7. a) Blood routine: ANC≥1.5×10^9/L, PLT≥80×10^9/L, Hb≥9.0 g/dL.Note: 14 days before the examination, it is not allowed to use any blood components, cell growth factors and other interventions to make the indicators reach the normal range；b) Liver function: TBIL≤ 1.5 times the upper limit of the normal value, ALB≥30 g/L, ALT and AST ≤ 2.5 times the upper limit of normal value; The value of patients with liver metastasis did not exceed 5 times the upper limit of normal value.; c) Renal function: Scr≤1.5 times the upper limit of the normal value,Ccr≥50mL/min (Cockcroft-Gault); d) Coagulation function is normal (PT and APPT are within 1.5 times of the upper limit of normal value);
8. Women of childbearing age had a negative pregnancy test result within 7 days before enrollment. Female subjects and their spouses received effective contraceptives during and within 6 months of treatment；
9. Weight≥40 kg；
10. Subjects with herpes in the reproductive organs needed three months after the end of herpes.
11. The informed consent was voluntarily signed and the expected compliance was good.

Exclusion Criteria:

1. Patients diagnosed with pancreatic cancer without pathology and/ or cytology;
2. The target lesion has received local non-drug therapy (including radiotherapy, physical and/or chemical ablation, etc.), and no imaging disease progression has occurred；
3. Central nervous system metastasis or cancerous meningitis is known to occur. For suspected central nervous system metastasis, head MRI examination is required;
4. Patients with Vater's ampullary carcinoma or biliary adenocarcinoma；
5. Patients with partial or complete intestinal obstruction and complete biliary obstruction that cannot be relieved by active treatment;
6. With more than a moderate amount of ascites, or after conservative medical treatment (such as diuresis, sodium restriction, excluding ascites drainage) for 2 weeks, the ascites still shows a progressive increase；
7. A history of other malignant tumors in the past 5 years, except for the following two cases: a. Other malignant tumors treated by a single operation, achieving 5 consecutive years of disease-free survival; b. Cured skin basal cell carcinoma and cured cervical carcinoma in situ;
8. Pregnant or lactating female;
9. Suffer from severe chronic or active infections, including tuberculosis, syphilis, AIDS (HIV antibody positive)；
10. Hypertension that cannot be effectively controlled (defined as systolic/diastolic blood pressure ≥150/100 mmHg or meeting one of them after treatment with standardized antihypertensive drugs); Angina pectoris or unstable angina pectoris occurred within the last 3 months, myocardial infarction or cardiac insufficiency occurred within 1 year before enrollment (heart function ≥ New York Heart Association NYHA grade II); Severe arrhythmia requiring medical treatment, left ventricular ejection fraction <50%; QTc interval male>450ms, female>470ms; Or there are risk factors for torsade de pointes ventricular tachycardia, such as clinically significant hypokalemia as judged by the investigator; Family history of long QT syndrome or family history of arrhythmia (such as WPW syndrome); Schizophrenia, or history of psychotropic drug abuse;
11. Suffer from acute or chronic active hepatitis (Hepatitis B reference: HbsAg positive and HBV DNA viral load ≥200IU/mL or ≥10^3 copies/mL, HCV antibody positive and HCV RNA positive);
12. Received any of the following treatments within a certain period of time before enrollment: a.Received second-level or above surgery within 4 weeks (regardless of tumor-related or not), except for minimally invasive surgery under gastrointestinal endoscope; b. Received extended-range radiotherapy within 4 weeks, or received local-range radiotherapy within 2 weeks; c. Other clinical studies have been taken in the past 4 weeks; d. Received local anti-tumor therapy within 4 weeks；
13. Toxicity caused by previous anti-tumor therapy before the first dose has not yet recovered to NCI CTCAE version 5.0 grade 0 or 1 (excluding hair loss, skin pigmentation, and non-clinically significant and asymptomatic laboratory abnormalities)；
14. Known to be allergic or intolerant to OH2 and its excipients；
15. The researchers believe that there is any reason why the patient is not suitable to participate in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
The objective response rate of patients with pancreatic cancer receiving OH2 injection. | 2 years
  Tumor evaluation is performed according to RECIST1.1 and iRECIST1.1. The assessment result is the number and proportion of subjects with complete response + partial response.

SECONDARY OUTCOMES:
Evaluation of safety of OH2 injection in patients with pancreatic cancer. | 2 years
  According to the version 5.0 of the National Cancer Institute Common Terminology Criteria for Adverse Events, the adverse events during the entire study period are evaluated.
The disease control rate of patients with pancreatic cancer receiving OH2 injection. | 2 years
  Tumor evaluation is performed according to RECIST1.1 and iRECIST1.1. The assessment result is the number and proportion of subjects with complete response + partial response + stable disease.
The duration of response of patients with pancreatic cancer receiving OH2 injection | 2 years
  Tumor evaluation is performed according to RECIST1.1 and iRECIST1.1. The time from the first assessment of complete response or partial response to the first assessment of disease progression or death from any cause.
The progression free survival of patients with pancreatic cancer receiving OH2 injection. | 2 years
  Tumor evaluation is performed according to RECIST1.1 and iRECIST1.1. Time from start of treatment to disease progression.
To evaluate the impact of OH2 in patients with pancreatic cancer on the quality of life | 2 years
  Evaluation based on EORTC QLQ-C30.

CONTACTS AND LOCATIONS:
Locations (1):
- Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality, China